CLINICAL TRIAL: NCT06591975
Title: Investigation of the Relationship Between Upper Extremity Function and Balance and Functional Mobility in Parkinson's Disease
Brief Title: The Relationship Between Upper Extremity Function and Balance and Functional Mobility in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, assistant professor, Cumhuriyet University
Other Study IDs: PD-hand-balance-mobility
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; upper extremity; balance; mobility
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individials with Parkinson's Disease: Parkinson's Disease patients will be included in this study. Inclusion and exclusion criteria will be considered.

SUMMARY:
Parkinson's Disease (PD) is the second most common neurodegenerative disease, affecting 2-3% of the population aged 65 and over, characterized by the loss of dopaminergic neurons. The basal ganglia play a significant role in the pathogenesis of PD. The lesions of the basal ganglia impair the ability of patients to perform complex, goal-oriented, and skill-requiring movements. Consequently, motor symptoms such as bradykinesia, rigidity, hypokinesia, and tremor, which are progressively worse, are added to the clinical picture of the disease.

These symptoms, which cause movement and activity limitations in individuals with PD, also affect upper extremity functions, balance, and functional mobility. Impairment of upper extremity functions, commonly seen from the early stages of the disease, can affect many basic activities of daily living, including buttoning clothes, tying shoelaces, sewing, writing, eating, and using various modern devices. Balance and mobility disorders are among the most debilitating features of the disease, as they lead to the deterioration of physical functions in PD. Balance and mobility issues in PD are identified as key determinants of the increasing fear of falling and the resulting decline in quality of life. Various factors such as rigidity, bradykinesia, impaired postural adjustments, and decreased sensory integration contribute to the negative impact on balance and mobility in individuals with PD.

Proper balance and mobility performance are achieved through synergistic control during both dynamic and static postures between proximal body segments such as the trunk, spine, and pelvis. This contributes to the mobility of distal segments and the functionality of the upper extremities. Additionally, the contribution of upper extremity functions to balance and mobility has been demonstrated in healthy populations. Current literature also reveals that treatment programs targeting the upper extremities can improve mobility and balance, especially in neurological patient populations.

In conclusion, balance and mobility disorders in Parkinson's disease can reduce proximal stability and affect hand dexterity. This study aims to examine the relationship between hand dexterity, balance, and functional mobility in individuals with PD.

DETAILED DESCRIPTION:
According to the sample size calculation, at least 26 diagnosed PD will be included. Participants' demographic characteristics will be taken initially and the stage will be recorded according to the Hoehn and Yahr Scale. Then, upper extremity functions, balance, and functional mobility will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having accepted participation in the study after being provided with detailed information about the research
* Having been diagnosed with only Parkinson's Disease by a specialist physician
* Having a Standardized Mini-Mental Test score greater than 24
* Being in stages 1 to 3 according to the Hoehn and Yahr Scale

Exclusion Criteria:

* Having any vision, hearing, or perceptual issues that could affect the research outcomes
* Having an orthopedic problem in the upper extremity that could impact hand dexterity, balance, or mobility
* Having a cardiovascular, pulmonary, or hormonal disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred with a diagnosis of Parkinson's Disease (PD) to the Department of Physiotherapy and Rehabilitation at the University by a specialist physician from the Department of Neurology at the University Medical Faculty Research and Application Hospital will be included in the study
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The Nine-Hole Peg Test | Assessment will be conducted immediately after enrollment.
  The Nine-Hole Peg Test (9-HPT) will be used to assess upper extremity functions. The 9-HPT evaluates hand dexterity based on performance. The test consists of nine pegs and nine holes (peg length: 32 mm, peg diameter: 7 mm, hole diameter: 7.5 mm, hole depth: 13 mm). In the test, the participant is asked to pick up the pegs one by one and place them into the holes as quickly as possible, and once all the pegs are placed, they are asked to collect them again without delay. The test begins with the command "start" and the test duration is recorded in seconds using a stopwatch. It is performed separately for both the right and left hands. The 9-HPT has been determined to be valid and reliable in individuals with Parkinson's Disease.
The Berg Balance Scale | Assessment will be conducted immediately after enrollment.
  The balance assessment will be conducted using the Berg Balance Scale (BBS). The BBS measures the ability to maintain balance during different positions, postural changes, and movements. It is widely used in Parkinson's Disease (PD) and is a highly reliable and valid scale. The scale consists of 14 tests, each rated on a 4-point scale. The highest score is 56; a score of 0-20 indicates balance impairment (high risk of falling), 21-40 suggests acceptable balance (moderate risk of falling), and 41-56 indicates good balance (low risk of falling). Lower scores point to a loss of static or dynamic balance during daily activities, indicating the presence of a higher risk of falls and functional limitations.
The Timed Up and Go Test | Assessment will be conducted immediately after enrollment.
  Functional mobility will be assessed using the Timed Up and Go Test (TUG). During the test, the individual is asked to rise from a chair, walk 3 meters, turn to the right or left, and then walk back to the chair at a brisk pace without running, and sit down again. The test begins with the command "go" and the time is recorded using a stopwatch. In our study, the TUG will be performed three times, and the best score will be used for analysis. The TUG has been found to be valid and reliable in individuals with Parkinson's Disease (PD).
The timed 360° turn test | Assessment will be conducted immediately after enrollment.
  The timed 360° turn test is an easily administered, not time-consuming, and specific measurement tool to assess turning ability. It measures the time taken for an individual to 360° turn around in a standing position. The timed 360° turn test is also correlated with balance and functional mobility.
Functional Reach Test | Assessment will be conducted immediately after enrollment.
  The Functional Reach Test assesses balance by measuring the limits while the patient reaches forwards as far as possible, having the arms in 90° flexion and without lifting the heels off the floor.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- [Background] Milosevic M, McConville KM, Masani K. Arm movement improves performance in clinical balance and mobility tests. Gait Posture. 2011 Mar;33(3):507-9. doi: 10.1016/j.gaitpost.2010.12.005. Epub 2011 Jan 11. PMID 21227695
- [Background] Kalkan AC, Kahraman T, Ugut BO, Colakoglu BD, Genc A. A comparison of the relationship between manual dexterity and postural control in young and older individuals with Parkinson's disease. J Clin Neurosci. 2020 May;75:89-93. doi: 10.1016/j.jocn.2020.03.018. Epub 2020 Mar 20. PMID 32201026